CLINICAL TRIAL: NCT06118684
Title: An Open-label, Healthy Subject, Two-part Study to Assess the Effect of Verapamil on Systemic Exposure of EP395 (Part A), and to Assess the Effect of EP395 on Systemic Exposure of Midazolam and Digoxin (Part B)
Brief Title: Clinical Trial to Assess Effect of Verapamil on Systemic Exposure of EP395 and Effect of EP395 on Systemic Exposure of Midazolam and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiEndo Pharmaceuticals (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP395-004
Record Dates: First submitted 2023-10-20; First posted 2023-11-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Verapamil; Midazolam; Digoxin

STUDY DESIGN:
Intervention Model Description: This is a single centre, open label trial to assess the impact of CYP3A4 and Pgp inhibition on the PK of EP395 (Part A); and, to assess the impact of EP395 on the PK of a CYP3A4 substrate and a Pgp substrate (Part B). Parts A and B of the trial may be conducted concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - EP395 as a 'victim' of DDIs (Experimental): Part A will investigate EP395 as a 'victim' of DDIs. The impact of CYP3A4 and P-glycoprotein (Pgp) inhibition on the pharmacokinetics (PK) of EP395 will be assessed. Verapamil has been selected as a moderate inhibitor of CYP3A4 and an inhibitor of Pgp.
  Interventions: Drug: EP395 (Part A and B); Drug: Verapamil (Part A)
- Part B - EP395 as a 'perpetrator' of DDIs (Experimental): Part B will investigate EP395 as a 'perpetrator' of DDIs. The impact of EP395 on the PK of a CYP3A4 substrate and a Pgp substrate will be assessed. Midazolam has been selected as the CYP3A4 substrate and digoxin as the Pgp substrate.
  Interventions: Drug: EP395 (Part A and B); Drug: Midazolam (Part B); Drug: Digoxin (Part B)

INTERVENTIONS:
Drug: EP395 (Part A and B) — EP395 (test product) oral capsule 125 mg. Part A: Dose: 1 capsule as a single dose on Day 1 and Day 14, total daily dose: 125 mg.
  Part B: Dose: 3 capsules once daily on Days 9 to 28, total daily dose: 375 mg.
Drug: Verapamil (Part A) — Verapamil (CYP3A4/Pgp inhibitor), tablet 40 mg. Part A: Dose: 3 tablets twice daily Days 10 to 18, total daily dose: 240 mg.
  Arms: Part A - EP395 as a 'victim' of DDIs
Drug: Midazolam (Part B) — Midazolam (CYP3A4 substrate) oral solution 1 mg/mL. Part B: Dose: 4 mL as a single dose on Day 1 and Day 24, total daily dose: 4 mg.
  Arms: Part B - EP395 as a 'perpetrator' of DDIs
Drug: Digoxin (Part B) — Digoxin (Pgp substrate) tablet 0.25 mg. Part B: Dose: 1 tablet as a single dose on Day 1 and Day 24, total daily dose: 0.25 mg.
  Arms: Part B - EP395 as a 'perpetrator' of DDIs

SUMMARY:
The aim of this trial is to assess the potential key drug-drug interactions with EP395 in the clinical setting.

DETAILED DESCRIPTION:
This is an open-label, healthy subject, two-part study to assess the effect of verapamil on systemic exposure of EP395 (Part A), and to assess the effect of EP395 on systemic exposure of midazolam and digoxin (Part B).

The overall aim of this trial is to assess the potential key drug-drug interactions (DDIs) with EP395 in the clinical setting. The trial will be in two parts:

Part A will investigate EP395 as a 'victim' of DDIs. The impact of CYP3A4 and P-glycoprotein (Pgp) inhibition on the pharmacokinetics (PK) of EP395 will be assessed. Verapamil has been selected as a moderate inhibitor of CYP3A4 and an inhibitor of Pgp.

Part B will investigate EP395 as a 'perpetrator' of DDIs. The impact of EP395 on the PK of a CYP3A4 substrate and a Pgp substrate will be assessed. Midazolam has been selected as the CYP3A4 substrate and digoxin as the Pgp substrate.

The trial population is healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand the information on the nature, the scope, and the relevance of the trial, and to provide voluntary, written informed consent to participate in the trial before any trial-related procedures.
2. Healthy male or female participant aged 18 to 55 years, inclusive.
3. Body mass index ≥ 19.0 and ≤ 33.0 kg/m2 at the time of the screening visit.
4. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.
5. Non-smoker, or former smoker with <10 pack years who stopped smoking (including e-cigarettes) at least 6 months before the screening visit.
6. Women of childbearing potential (WOCBP) must:

   1. have a negative pregnancy test (blood) at the screening visit and (urine) Day 1.
   2. agree to use, and be able to comply with, highly effective measures of contraceptive control (failure rate less than 1% per year when used consistently and correctly) without interruption, during trial participation and until 90 days after the last IMP intake.
   3. agree to abstain from breast feeding during the trial participation and for 90 days after the last IP intake.

Women defined as of non-childbearing potential are postmenopausal (no menses for at least 1 year without alternative medical cause [follicle stimulating hormone, FSH, measurement in serum may be done as additional confirmation at Investigator's discretion]) or surgically sterile women (tubal ligation, hysterectomy, or bilateral oophorectomy).

Men must agree to use a condom during sexual intercourse with WOCBP during treatment and for 90 days after the last IP intake and should not donate sperm during this time.

Exclusion Criteria:

Participants must not enter the trial if any of the following exclusion criteria are fulfilled:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results, or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the (first) administration of IMP.
3. Presence or history of lung disease, e.g., asthma, chronic obstructive pulmonary disease.
4. Presence or history of significant gastrointestinal medical condition that could lead to abnormal absorption.
5. History of or active tuberculosis at the time of the screening visit based on participant anamnesis. Participants who have been living together with another person with active tuberculosis at any time over the past 10 years will also be excluded.
6. Clinically significant abnormality on 12-lead ECG at the screening visit or Day 1 pre-dose, including prolonged QTcF (>450 msec men or >470 msec women) or PR interval >210 msec.
7. Abnormal renal function at the time of the screening visit:

   * serum creatinine >upper limit of normal (ULN); and/or
   * estimated glomerular filtration rate <60 mL/min according to the revised Lund-Malmö GFR estimating equation.
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 x ULN at the time of the screening visit.
9. Use of prescription or non-prescription medications or herbal remedies within 28 days prior to Day 1, or unable to refrain from prescription or non-prescription medications or herbal remedies during the trial, with the following exceptions:

   * hormone replacement therapy (HRT)
   * contraception
   * occasional use of paracetamol Note: other medications will be reviewed by the Medical Monitor and a participant may be included if both the Investigator and Medical Monitor agree that the medication will not interfere with the trial assessments or participant's safety.
10. Live vaccine within 28 days or any other vaccine within 14 days prior to Day 1 until 28 days after the final dose (with the exception of COVID-19 vaccine boosters).
11. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
12. Positive screening result for drugs of abuse, cotinine or alcohol at the screening visit or on admission to the trial site prior to the (first) administration of the IMP. A positive urine cotinine test (≥200 ng/mL) at screening or at Day -1 will exclude the participant from trial participation.
13. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
14. Presence or history of drug abuse, as judged by the Investigator.
15. History of, or current use of anabolic steroids, as judged by the Investigator.
16. Excessive caffeine consumption defined by a daily intake of > 5 cups (1 cup = approximately 240 mL) of coffee, or equal amount in other caffeine containing beverages, or unable to refrain from caffeine containing beverages, including energy drinks, during the trial, as judged by the Investigator.
17. Former smoker with >10 pack years, or smoking (including use of e-cigarettes and vapes) within 6 months of the screening visit, or unable to refrain from smoking throughout the trial.
18. Use of nicotine replacement products within 2 weeks of the screening visit and unable to refrain from nicotine replacement products throughout the trial.
19. Participants who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
20. Known hypersensitivity to macrolides or EP395 or any of the excipients (dicalcium phosphate, croscarmellose sodium, magnesium stearate, microcrystalline cellulose).
21. History of hypersensitivity to or contraindication (as indicated in the SmPC) to verapamil (Part A) or digoxin and/or midazolam (Part B).
22. Any clinically significant allergy, as judged by the Investigator.
23. Planned treatment or treatment with another investigational drug within 5 half-lives of said drug or 3 months prior to first IMP administration, whichever is longer. Participants consented and screened, but not dosed in previous Phase 1 trials are not excluded.
24. Employees of the Sponsor or employees or relatives of the Investigator.
25. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the last three months prior to the first IMP administration.
26. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Part A: PK parameters of EP395 - AUC0-24 | Days 1 to 6 and Day 14 to 19
  Area under the plasma concentration vs. time curve from timepoint 0 to 24 hours of EP395.
Part A: PK parameters of EP395 - AUC0-inf | Days 1 to 6 and Day 14 to 19
  Area under the plasma concentration vs. time curve from timepoint 0 to infinity of EP395.
Part A: PK parameters of EP395 - AUC%extrap | Days 1 to 6 and Day 14 to 19
  Percent of AUCinf derived from extrapolation of the plasma concentration vs. time curve of EP395.
Part A: PK parameters of EP395 - CL/F | Days 1 to 6 and Day 14 to 19
  Apparent total body clearance following extravascular administration of EP395.
Part A: PK parameters of EP395 - Cmax | Days 1 to 6 and Day 14 to 19
  Maximum observed plasma concentration of EP395.
Part A: PK parameters of EP395 - Tmax | Days 1 to 6 and Day 14 to 19
  Time to occurrence of Cmax of EP395.
Part A: PK parameters of EP395 - T1/2 | Days 1 to 6 and Day 14 to 19
  Terminal elimination half-life of EP395.
Part A: PK parameters of EP395 - Vz/F | Days 1 to 6 and Day 14 to 19
  Volume of distribution following extravascular administration of EP395.
Part B: PK parameters of midazolam and digoxin - AUC0-24 | Days 1 to 3/6 and Day 24 to 29
  Area under the plasma concentration vs. time curve from timepoint 0 to 24 hours of midazolam and digoxin.
Part B: PK parameters of midazolam and digoxin - AUC0-inf | Days 1 to 3/6 and Day 24 to 29
  Area under the plasma concentration vs. time curve from timepoint 0 to infinity of midazolam and digoxin.
Part B: PK parameters of midazolam and digoxin - AUC%extrap | Days 1 to 3/6 and Day 24 to 29
  Percent of AUCinf derived from extrapolation of the plasma concentration vs. time curve of midazolam and digoxin.
Part B: PK parameters of midazolam and digoxin - Cmax | Days 1 to 3/6 and Day 24 to 29
  Maximum observed plasma concentration of midazolam and digoxin.
Part B: PK parameters of midazolam and digoxin - Tmax | Days 1 to 3/6 and Day 24 to 29
  Time to occurrence of Cmax of midazolam and digoxin.
Part B: PK parameters of midazolam and digoxin - T1/2 | Days 1 to 3/6 and Day 24 to 29
  Terminal elimination half-life of midazolam and digoxin.

SECONDARY OUTCOMES:
Part A: Assessment of adverse event occurrence | From screening to Day 30.
Part A: Absolute change from baseline in vital signs (Systolic and diastolic blood pressure) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant.
Part A: Absolute change from baseline in vital signs (Pulse) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant.
Part A: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (heart rate) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting heart rate (HR) will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part A: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (PQ/PR interval) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting PQ/PR interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part A: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QRS interval) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QRS interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part A: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QT interval) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QT interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part A: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QTcF interval) | Screening (Day -28 to Day -1), Day 1, Day 10-19
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QTcF interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part A: Absolute change from baseline in safety laboratory analytes (haematology). | Screening (Day -28 to Day -1), Day -1, Day 10, Day 14, Day 19
  Erythrocyte count, Leukocyte count with differential count, Haematocrit (EVF), Haemoglobin (Hb), Mean corpuscular haemoglobin (MCH), Mean corpuscular volume (MCV), Platelet count.
  Absolute changes from baseline will be summarized for all assessed time points.
Part A: Absolute change from baseline in safety laboratory analytes (clinical chemistry). | Screening (Day -28 to Day -1), Day -1, Day 10, Day 14, Day 19
  Alanine aminotransferase (ALT), Albumin, Alkaline phosphatase (ALP), Aspartate aminotransferase (AST), Bilirubin (total and conjugated), Calcium, Creatinine (estimated Glomerular Filtration Rate [eGFR] included), Gamma glutamyl transferase, Glucose (non-fasting, at screening only), Lactate dehydrogenase, Phosphate, Potassium, Protein (total), Sodium, Urea
  Absolute changes from baseline will be summarized for all assessed time points.
Part A: Absolute change from baseline in safety laboratory analytes (coagulation). | Screening (Day -28 to Day -1), Day -1, Day 10, Day 14, Day 19
  Activated Partial Thromboplastin Time (APTT), Prothrombin Complex International Normalised Ratio (PK[INR])
  Absolute changes from baseline will be summarized for all assessed time points.
Part B: Assessment of adverse event occurrence | From screening to Day 30.
Part B: Absolute change from baseline in vital signs (Systolic and diastolic blood pressure) | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant.
Part B: Absolute change from baseline in vital signs (Pulse) | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (heart rate). | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting heart rate (HR) will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (PQ/PRinterval). | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting PQ/PR interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QRS interval). | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QRS interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QT interval). | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QT interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters (QTcF interval). | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting QTcF interval will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in 12-lead Electrocardiogram (ECG) parameters | Screening (Day -28 to Day -1), Day 1, Day 9, Day 16, Day 24, Day 28
  Number of patients with any clinically significant change in 12-lead Electrocardiogram (ECG) parameters.
  The resting heart rate (HR) and PQ/PR, QRS, QT and QTcF intervals will be recorded. Any abnormalities in ECG will be specified and documented as clinically significant or not clinically significant.
Part B: Absolute change from baseline in safety laboratory analytes (haematology). | Screening (Day -28 to Day -1), Day -1, Day 9, Day 16, Day 23, D28
  Erythrocyte count, Leukocyte count with differential count, Haematocrit (EVF), Haemoglobin (Hb), Mean corpuscular haemoglobin (MCH), Mean corpuscular volume (MCV), Platelet count.
  Absolute changes from baseline will be summarized for all assessed time points.
Part B: Absolute change from baseline in safety laboratory analytes (clinical chemistry). | Screening (Day -28 to Day -1), Day -1, Day 9, Day 16, Day 23, D28
  Alanine aminotransferase (ALT), Albumin, Alkaline phosphatase (ALP), Aspartate aminotransferase (AST), Bilirubin (total and conjugated), Calcium, Creatinine (estimated Glomerular Filtration Rate [eGFR] included), Gamma glutamyl transferase, Glucose (non-fasting, at screening only), Lactate dehydrogenase, Phosphate, Potassium, Protein (total), Sodium, Urea
  Absolute changes from baseline will be summarized for all assessed time points.
Part B: Absolute change from baseline in safety laboratory analytes (coagulation). | Screening (Day -28 to Day -1), Day -1, Day 9, Day 16, Day 23, D28
  Activated Partial Thromboplastin Time (APTT), Prothrombin Complex International Normalised Ratio (PK[INR])
  Absolute changes from baseline will be summarized for all assessed time points.
Part B: PK parameters of EP395 and its major metabolites (Cmax) | Days 1 to 3/6 and Day 24 to 29
  The ratios of EP395 metabolite to parent systemic exposures in terms of Cmax and AUC0-24 will be calculated and expressed as percentages.
Part B: PK parameters of EP395 and its major metabolites (AUC0-24) | Days 1 to 3/6 and Day 24 to 29
  The ratios of EP395 metabolite to parent systemic exposures in terms of Cmax and AUC0-24 will be calculated and expressed as percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Schultze, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No